CLINICAL TRIAL: NCT07194473
Title: ZeroOCD: Learn to Overcome Contamination OCD With Your Smartphone: An Augmented Reality Cognitive Behavioral Therapy App for Obsessive-Compulsive Disorder: Randomized Controlled Trial
Brief Title: ZeroOCD: Learn to Overcome Contamination OCD With Your Smartphone
Acronym: ZeroOCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: University of Bern (Other); Stockholm University (Other); Thomas More University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Tara Donker, Associate Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZeroOCD/FP-1478
Record Dates: First submitted 2025-09-03; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Obsessive Compulsive Disorder; Augmented Reality; Smartphone; Randomized Controlled Trial; Cost-effectiveness
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZeroOCD AR-CBT App + 3 therapist support sessions (Experimental): Participants will use the ZeroOCD smartphone application, which delivers 9 modules of augmented reality exposure therapy and cognitive behavioral therapy principles. This group will also receive 3 videoconferencing sessions with a therapist at the beginning, middle, and end of the 10-week treatment period.
  Interventions: Behavioral: ZeroOCD
- Videoconferencing CBT (Active Comparator): Participants will receive 9 weekly sessions of manualized Cognitive Behavioral Therapy with Exposure and Response Prevention (ERP) delivered via videoconferencing by trained therapists.
  Interventions: Behavioral: Videoconferencing CBT
- Waitlist control group (No Intervention): Participants in this group will receive access to the ZeroOCD app with therapist support on request after a 10-week waiting period.

INTERVENTIONS:
Behavioral: ZeroOCD — The ZeroOCD app contains the following components:
  psychoeducation, detecting obsessive thoughts, coping with obsessions, goal setting, fear curve explanation, exposure with AR, re-exposure with AR, exposure hierarchy, exposure in real-life, re-exposure in real life and relapse prevention
  Other Names: ZeroOCD AR-CBT App + 3 therapist support sessions
  Arms: ZeroOCD AR-CBT App + 3 therapist support sessions
Behavioral: Videoconferencing CBT — Videoconferencing CBT contains the following chapters:
  psychoeducation, detecting obsessive thoughts, coping with obsessions, goal setting, fear curve explanation, exposure hierarchy, exposure in real-life, re-exposure in real life and relapse prevention
  Arms: Videoconferencing CBT

SUMMARY:
This study is a three-arm randomized controlled trial designed to evaluate the efficacy of a smartphone-based augmented reality (AR) cognitive behavioral therapy (CBT) app, called ZeroOCD, for individuals with elevated contamination-related obsessive-compulsive disorder (OCD) symptoms. The AR-CBT app will be compared to both an active control condition (manualized CBT via videoconferencing) and a waitlist control group.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a prevalent and disabling condition, with contamination fears being one of its most common presentations. While Cognitive-Behavioral Therapy (CBT) with Exposure and Response Prevention (ERP) is a first-line treatment, many individuals face barriers to accessing it, such as cost, stigma, and availability of therapists. This multicenter trial, conducted in the Netherlands, Belgium, Sweden, and Switzerland, will recruit a total of 189 individuals experiencing contamination-related obsessive-compulsive symptoms. Participants will be randomized to one of three study conditions (allocation ratio 2:2:1): The first group (n = 75) receives access to ZeroOCD, an augmented reality (AR) based smartphone application, which provides CBT and ERP for contamination fears, along with three therapist support sessions via videoconferencing. The second group (n = 75) receives weekly CBT for OCD via videoconferencing (nine sessions in total). The third group is a waitlist control group (n = 39), who will receive access to the smartphone application with minimal therapist support on request after 10 weeks in the study. The study aims to evaluate the effectiveness of the ZeroOCD intervention compared to both a waitlist control and videoconferencing CBT, and to assess cost-effectiveness and usability. Assessments are conducted at baseline, 10 weeks post-randomization, and at 6-month follow-up for the intervention groups. Participants in the waitlist group complete assessments at baseline, 10 weeks post-randomization, and receive access to the ZeroOCD intervention 10 weeks after randomization. Further, the waitlist group will complete an assessment 20 weeks post-randomization. The study is a multicenter trial involving participants in Switzerland, the Netherlands, Belgium, and Sweden.

ELIGIBILITY:
Inclusion Criteria:

* • OCD symptoms, mean score > 7 on the Yale Brown Obsessive Compulsive Scale (Y-BOCS)

  * Fear of contamination OCD symptoms, mean score > 6 on the Padua Inventory contamination fear subscale (PI)
  * Having access to a compatible smartphone
  * Having an internet connection
  * Proficiency in one of the countries' languages (i.e., Dutch/ Flemish, German, or Swedish)
  * Willing to participate in the research study and provide informed consent

Exclusion Criteria:

* • Having been diagnosed with bipolar or psychotic disorder (self-report)

  * Severe depressive symptoms (Patient Health Questionnaire, PHQ-9, score > 20)
  * Reporting suicidality (PHQ-9, item 9 > 2 points at screening)
  * Fear of contamination due to disorder other than OCD (clinical judgment based on results from the Yale Brown Obsessive Compulsive Scale, Y-BOCS, Generalized Anxiety Disorder-7 items, GAD-7, Short Health Anxiety Inventory, SHAI)
  * Parallel psychological treatment
  * Non-stable dosage of psychoactive medication during the last three months or planned changes during the study period.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-09-21 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
OCD Symptoms (Interview) | At baseline, At 10 weeks, At 20 weeks (only WL condition) At 24 weeks
  Yale-Brown Obsessive Compulsive Scale (Y-BOCS): Change from baseline in the observer-rated severity of OCD symptoms. This is a 10-item, clinician-rated scale that provides separate subtotals for the severity of obsessions and compulsions. Total scores range from 0 to 40, with higher scores indicating more severe symptoms. The Y-BOCS is also used for the eligibility (mean score > 7).

SECONDARY OUTCOMES:
OCD symptoms (Self-report) | At baseline, During treatment (every week) At 10 weeks, At 24 weeks
  4-item Obsessive-Compulsive Inventory (OCI-4): Change from baseline in the self-reported OCD symptom severity. This shorter form of the OCI-R consists of 4 Items that quantify the symptom severity related to OCD. Each item is rated on a scale from 0 to 4, with total scores ranging from 0 to 16, with higher scores indicating more severe symptoms.
Fear of Contamination | At baseline, At 10 weeks, At 20 weeks (only WL condition) At 24 weeks
  Padua Inventory (PI) Contamination Fear Subscale: Change from baseline in the self-reported fear of contamination. This is a 10-item subscale that quantifies the severity of contamination-related obsessions, with each item rated on a 5-point Likert scale. A score of 6 or higher on this scale is an inclusion criterion for the study. The PI is also used for the eligibility (mean score > 6).
Depression | At baseline, At 10 weeks, At 24 weeks
  Patient Health Questionnaire-9 (PHQ-9): Change from baseline in self-reported depressive symptom severity. This is a 9-item measure where each item corresponds to a DSM-5 criterion for major depression. Scores range from 0 to 27, and a score of >20 is an exclusion criterion. The PHQ-9 is also used for the eligibility (severe depressive symptoms: score > 20; suicidality: item 9 score > 2).
Anxiety | At baseline, At 10 weeks, At 24 weeks
  Generalized Anxiety Disorder 7-item scale (GAD-7): Change from baseline in self-reported anxiety symptom severity. This is a 7-item measure with scores ranging from 0 to 21. It will also be used at baseline to help determine if contamination fears are due to GAD rather than OCD.
Current Distress/Disgust | up to ten weeks
  Subjective Units of Distress Scale (SUDS): Measurement of current distress and disgust levels before, during, and after exposure tasks within the ZeroOCD app. This is an ecological momentary assessment (EMA) where participants rate their distress on a visual analog scale from 0 to 10.
Social Functioning | At baseline, At 10 weeks, At 24 weeks
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0): Change from baseline in self-reported general functioning and disability. This is a 36-item measure that evaluates functioning across six major life domains (e.g., cognition, mobility, life activities).
Health Related Quality of Life | At baseline, At 10 weeks, At 24 weeks
  EQ-5D-5L measures change from baseline in self-reported health-related quality of life. This is a 5-item standardized questionnaire that evaluates health status across five domains (e.g., mobility, self-care, pain/discomfort).
Societal Costs of a Treatment | At baseline, At 10 weeks, At 24 weeks
  Treatment Inventory of Costs in Patients with Psychiatric Disorders (TiC-P): Change from baseline in the utilization of healthcare services and productivity losses. This is a 36-item self-report measure used for the cost-effectiveness analysis.
Usability | At 10 weeks (only ZeroOCD condition), At 20 weeks (only WL condition)
  System Usability Scale (SUS): A global assessment of the subjective usability of the ZeroOCD app, measured post-treatment. This is a 10-item questionnaire with total scores ranging from 0 to 100, where higher scores indicate greater perceived usability.
Treatment Satisfaction | At 10 weeks (only intervention groups)
  Client Satisfaction Questionnaire (CSQ): A measure of client satisfaction with the received treatment, assessed post-treatment. This is an 8-item self-report measure with total scores ranging from 8 to 32, where higher scores indicate greater satisfaction.
Realism of AR-Environment | At 10 weeks (only ZeroOCD condition)
  Realism subscale of the IGroup Presence Questionnaire (IPQ): A measure to assess the perceived realism of the augmented reality (AR) environment, administered post-treatment to the ZeroOCD group. This is a 4-item subscale relevant for AR with each item assessed on a 7-point Likert scale (from -3 to 3).
Negative Effects of Treatment | At 10 weeks (only ZeroOCD and CBT condition), at 20 weeks (only waitlist condition)
  Negative Effects Questionnaire (NEQ): A measure to evaluate any negative effects of the psychological treatments, assessed at post-treatment and follow-up. This is a 20-item questionnaire where participants report on the occurrence, negative impact, and attributed cause of potential negative events.
Usage Data | up to ten weeks (only ZeroOCD and waitlist condition)
  To understand the dose-response relationship in treatment effectiveness by analyzing how participants interact with the ZeroOCD app. This involves collecting data automatically from the app for participants in the intervention condition. Data points include the frequency and duration of practice during AR exposure, time spent in each module, number of modules and pages completed, and number of log-ins.

OTHER OUTCOMES:
Reasons for discontinuation | up to ten weeks
  Reasons for discontinuation: to understand why participants stop with the treatment before the end of the treatment
Socio-demographic information | At baseline
  Socio-demographic questionnaire: To gather participant characteristics and demographics at the start of the study. This questionnaire collects information about participants' age, gender, education level, marital status, employment status, and treatment preference. It also gathers information on current or past psychological treatment and medication to confirm eligibility.
Health Anxiety | At baseline
  Short Health Anxiety Inventory (SHAI): A self-report measure to assess the presence of health anxiety at baseline, which is an exclusion criterion if judged to be the primary driver of contamination fears. This is an 18-item measure rated on a scale from 0 to 3.

CONTACTS AND LOCATIONS:
Locations (4):
- Thomas More Mechelen, Mechelen, Belgium
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands
- Stockholm University, Stockholm, Sweden
- UBERN, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code